CLINICAL TRIAL: NCT02345603
Title: Pilot Study of of Renal Arterial Sympathetic Denervation by Cryotherapy During Open Surgery for Aortic Aneurysm
Brief Title: Pilot Study of of Renal Arterial Sympathetic Denervation by Cryotherapy
Acronym: PRASDEN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, MD PhD professor Head of internal medicine, University Hospital, Linkoeping
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/45-31
Record Dates: First submitted 2014-12-18; First posted 2015-01-26 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryo-therapy (Experimental): Cryo-therapy of renal arteries
  Interventions: Procedure: Cryo-therapy
- Control (No Intervention): No intervention in renal arteries

INTERVENTIONS:
Procedure: Cryo-therapy — Cryo-therapy for about 60 seconds applied circumpherentially to each renal artery
  Arms: Cryo-therapy

SUMMARY:
Non-randomized study of 5 subjects that have been selected for prophylactic open surgery due to abdominal aortic aneurysm. During surgery the renal arteries are identified and subjected to about 60 seconds each of freezing by application of liquid nitrogen in dedicated catheters around the circumference of each artery. Another 5 patients that are not subjected to the freeze therapy serve as controls. Main outcome is change in ambulatory blood pressure levels.

DETAILED DESCRIPTION:
Non-randomized study of 5 subjects that have been selected for prophylactic open surgery due to abdominal aortic aneurysm. During the surgery the renal arteries at both sides are identified and subjected to about 60 seconds each of freezing by application of liquid nitrogen in dedicated catheters around the circumference of each artery. Renal arterial blood flow is checked by Doppler after the freezing procedure, during the surgery. Another 5 patients that are not subjected to the freeze therapy serve as controls. Main outcome is change in 24h ambulatory blood pressure levels and of course safety parameters such as creatinine levels.

ELIGIBILITY:
Inclusion Criteria:

* planned prophylactic surgery for abdominal aortic aneurysm

Exclusion Criteria:

* hypotension,
* inability to understand study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure levels | 2 months
  24 hour mean ambulatory blood pressure levels before and 2 months after surgery

SECONDARY OUTCOMES:
Levels of epinephrine and nor-epinephrine in urine | before and 2 months after surgery
  Collection of urine for analyses of stress hormones

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Linkoping, Linköping, Sweden